CLINICAL TRIAL: NCT04523077
Title: Association of Oral Lichen Planus and Thyroid Disease
Status: Completed | Type: Observational
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Božana Lončar Brzak, Assistant Professor, University of Zagreb
Other Study IDs: 01122019
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Oral Lichen Planus; Thyroid Diseases
Keywords: oral lichen planus; thyroid diseases
MeSH Terms: conditions — Lichen Planus, Oral; Thyroid Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oral lichen planus: Female patients of the Department of Oral Medicine with oral lichen planus
  Interventions: Diagnostic Test: determination of thyroid hormones and antibodies
- Control: Female patients of the Department of Oral Medicine without oral lichen planus or other immune disorders
  Interventions: Diagnostic Test: determination of thyroid hormones and antibodies

INTERVENTIONS:
Diagnostic Test: determination of thyroid hormones and antibodies — TSH, fT3, fT4, anti-TPO and anti-Tg were determined from blood sample

SUMMARY:
Thyroid disease is a common endocrine disorder. Oral lichen planus (OLP) is a chronic autoimmune disease that occurs on the oral mucosa in 1-2% of the general population.The purpose of this study was to determine whether there is an association between thyroid disease and oral planus lichen in the population of our patients. In the last few years, a couple of studies have been published in the world literature that have studied the possible association of these diagnoses in different populations. Most of the results showed a higher prevalence of thyroid disease in the population of lichen patients, compared with patients without lichen, although some results are contradictory. Some authors believe that the onset of OLP precedes thyroid dysfunction. In the population of Croatian patients with lichen, no research has been done to study the possible connection between these two diseases. The obtained results could help clarify whether there is a connection between these two diagnoses in the population of our lichen patients and enable earlier detection of patients with thyroid hypofunction.

ELIGIBILITY:
Inclusion Criteria:

* for test group: female patients of the Department of Oral Medicine School of Dental Medicine University of Zagreb with clinically and histopathologically confirmed oral lichen planus
* for control group: female patients of the Department of Oral Medicine School of Dental Medicine University of Zagreb, without oral lichen planus or other immune disorders; age matched to test group

Exclusion Criteria:

* male patients; female patients with immune disorders; female patients which are not age-matched to test group

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Oral lichen planus and thyroid diseases are more frequent in female gender. We wanted the groups to be as similar in characteristics as possible so we included only females.
Study Population: The study included female patients of the Department of Oral Medicine, age matched, with oral lichen planus and without oral lichen planus or other immune disorders. All patients included in the study made blood test and the results were analyzed with statistical methods.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
The prevalence of thyroid diseases in patients with oral lichen planus | January 2020-April 2020
  to determine whether there is a higher prevalence of thyroid disease in patients with oral lichen

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dental Medicine, University of Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Undecided